CLINICAL TRIAL: NCT05376670
Title: Patient Satisfaction and Long-term Safety of Intravesical Aminoglycoside Instillations in UTI Prevention
Acronym: INSTILMENT
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Manu Bilsen, MD, MD, PhD student, Department of Infectious Diseases, Principle Investigator, Leiden University Medical Center
Other Study IDs: nWMODIV2_2022013
Record Dates: First submitted 2022-04-28; First posted 2022-05-17 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Urinary Tract Infections; Recurrent Urinary Tract Infection
Keywords: Intravesical treatment
MeSH Terms: conditions — Urinary Tract Infections | interventions — Tobramycin; Amikacin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Intravesical aminoglycoside instillations — Overnight instillation of an aminoglycoside (CIC), varying treatment regimens
  Other Names: Intravesical gentamicin, tobramycin or amikacin

SUMMARY:
Antimicrobial prophylactic treatment of recurrent UTI is limited by emerging resistance, antibiotic allergies and intolerances. Intravesical aminoglycoside instillations (IAI) have been shown to reduce recurrence rate, without a short-term decline in kidney function or hearing. Thus far, treatment satisfaction has not yet been assessed, while this may play an important role in treatment adherence and persistence. Moreover, there is no data on the long-term safety of IAI, e.g. regarding the development of (pre)malignant bladder lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Currently receiving or having received (no minimal duration) continuous or post-coital IAI (gentamicin, tobramycin or amikacin) for recurrent UTI prophylaxis and treatment

Exclusion Criteria:

* Exclusively receiving IAI for 'on-demand' treatment of UTI and not prophylactic purposes
* Receiving IAI as suppressive therapy for chronic prostatitis
* Presence of a chronic indwelling catheter
* Patient has objected to the use of his/her data
* Inability to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include adult male and female patients receiving IAI for recurrent UTI at the infectious diseases outpatient clinic of the Leiden University Medical Centre. A proportion of study participants will have urological and/or neurological comorbidities and a history of other prophylactic treatments for recurrent UTI.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction regarding intravesical aminoglycoside instillations (IAI) | 1 year
  Measured with Treatment Satisfaction Questionnaire for Medication version II (TSQM-II), value ranging from 0 to 100 (with a score of 100 indicating the highest treatment satisfaction)

SECONDARY OUTCOMES:
Time to first UTI recurrence after initiation of IAI | First 6 months of IAI
Number of UTI recurrences | First 6 months of IAI
Number of UTI recurrences that are treated with IAI alone (no systemic antimicrobial therapy) | First 6 months of IAI
Number of patients that wish to (dis)continue IAI | 6 months after initiation of IAI
Proportion of patients that have a UTI episode caused by the same MDRO uropathogen as before start of IAI | 6 months after initiation of IAI

CONTACTS AND LOCATIONS:
Overall Officials: Manu Bilsen, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided